CLINICAL TRIAL: NCT02719847
Title: Additive Value of EBUS TBNA for Staging Non-Small Cell Lung Cancer in Patients Evaluated for Stereotactic Body Radiation Therapy
Brief Title: EBUS TBNA After PET/CT in Diagnosing Patients With Stage I-IIA Non-small Cell Lung Cancer Evaluated for Stereotactic Body Radiation Therapy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0615; NCI-2016-00571 (Registry Identifier: NCI CTRP Clinical Trial Registry)
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Non-Small Cell Lung; NSCLC; Suspected non small cell lung cancer; Endobronchial ultrasound-guided transbronchial needle aspiration; EBUS-TBNA
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- EBUS-TBNA: Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) performed after PET/CT, and before participant receives stereotactic body radiation therapy (SBRT). EBUS-TBNA results compared with the results of PET/CT.
  A conventional flexible bronchoscopy performed to examine the tracheobronchial tree, followed by a systematic examination of the accessible intra-thoracic lymph nodes using a linear array ultrasound bronchoscope.
  Interventions: Procedure: Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA)

INTERVENTIONS:
Procedure: Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) — Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) performed after PET/CT, and before participant receives stereotactic body radiation therapy (SBRT). EBUS-TBNA results compared with the results of PET/CT.

SUMMARY:
This clinical trial studies how well endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) after positron emission tomography/computed tomography (PET/CT) scan works in diagnosing patients with stage I-IIA non-small cell lung cancer evaluated for stereotactic body radiation therapy (SBRT). Performing EBUS-TBNA after PET/CT scan may help doctors learn more about the accuracy and ways to find early stage lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the use of EBUS-TBNA after a PET/CT as a means of improving the accuracy of lymph node staging in patients considered for SBRT.

SECONDARY OBJECTIVES:

I. To assess the usefulness of PET/CT as a diagnostic test in identifying N1 versus N0 staging.

II. To compare survival and recurrence rates in patients with discordant PET/CT and EBUS-TBNA.

III. To describe EBUS-TBNA and SBRT related complications.

OUTLINE:

Patients undergo EBUS-TBNA before SBRT.

After completion of study, patients are followed up at 6 weeks, then every 3 months for the first 2 years then twice a year for the following 3 years, and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be > 18 years old
2. Patient must have proven or suspected non small cell lung cancer (NSCLC) and be clinical Stage I or IIa, according to the 7th edition staging system of the American Joint Commission on Cancer for lung cancer (T1 or T2a, N0 or N1, M0)
3. Patient must have a PET/CT obtained within 40 days of having the EBUS-TBNA
4. Patient is being considered for SBRT
5. Patient or the patient's legally authorized representative must provide written informed consent prior to registration and any study-related procedures
6. If the patient is a survivor of a prior invasive cancer, all of the following criteria must apply: a) Patient has undergone potentially curative therapy for all prior malignancies b) No evidence of active / recurrent disease within 5 years

Exclusion Criteria:

1. Patient has received prior chemotherapy or radiotherapy for this cancer
2. Patients already scheduled to receive conventional radiotherapy, chemotherapy, biological therapy, vaccine therapy, or surgery as treatment (except at disease progression)
3. Patients malignancy is consistent with well differentiated neuroendocrine (carcinoid) histology
4. Patients who are planning to undergo treatment in a different institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-03-18 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Lymphnode Staging Accuracy | 1 day
  The use of EBUS-TBNA after a PET/CT as a means of improving the accuracy of lymphnode staging in patients considered for SBRT estimated as the proportion of patients identified concordantly as having N0 disease with both PET/CT and EBUS-TBNA.

CONTACTS AND LOCATIONS:
Overall Officials: George A. Eapen, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT02719847/ICF_000.pdf